CLINICAL TRIAL: NCT05160389
Title: A Single-Dose, Open-Label, Randomized, Three-Way, Crossover Study to Assess the Effect of Food on the Absorption and Bioavailability of PBI-200 in Normal Healthy Volunteers
Brief Title: A Study to Assess the Effect of Food on the Absorption and Bioavailability of PBI-200
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pyramid Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PBI-200-103
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Food Effect in Healthy Volunteers
Keywords: Volunteer

STUDY DESIGN:
Intervention Model Description: Single-dose, open-label, randomized, three-way crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fasted (Experimental): Study drug will be administered with water, after an overnight fast.
  Interventions: Drug: PBI-200
- Low-fat Meal (Experimental): Study drug will be administered with water, after an overnight fast, after which time a standard low-fat breakfast will be given.
  Interventions: Drug: PBI-200
- High-fat Meal (Experimental): Study drug will be administered with water, after an overnight fast, after which time a standard high-fat breakfast will be given.
  Interventions: Drug: PBI-200

INTERVENTIONS:
Drug: PBI-200 — Single dose of PBI-200

SUMMARY:
This is a single-dose, open-label, randomized, three-way crossover study to assess the effect of food on the absorption and bioavailability of PBI-200.

DETAILED DESCRIPTION:
This is a single-dose, open-label, randomized, three-way crossover study to assess the effect of food on the absorption and bioavailability of PBI-200, administered orally under fasted and fed conditions.

The study will enroll 18 healthy adult volunteers to ensure study completion of at least 12 evaluable volunteers. The study will be conducted in 3 groups, with each group enrolling 6 volunteers. As this is a crossover study, each volunteer will serve as their own control.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or non-pregnant, non-lactating female between 18 and 55 years of age (inclusive).
* Body Mass Index (BMI) between 18 and 32 kg/m² (inclusive).
* Non-smoking/non-vaping, healthy, with no history of clinically relevant medical illness.

Key Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, respiratory, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease which, in the opinion of the Investigator, would jeopardize the safety of the volunteer or impact the validity of the study results.
* History of gastrointestinal/hepatobiliary or other surgery that may affect PK profiles (i.e., hepatectomy, gastric, bypass, or digestive organ resection).
* Intolerance to repeated venipuncture.
* Smoking or use of tobacco products (including vaping) within 3 months prior to the first study drug administration.
* Have a positive drug/alcohol screen, or history or presence of alcoholism or drug abuse within 6 months of first study drug administration.
* Volunteers with a corrected QT using Fredericia's formula (QTcF) prolongation over 450 milliseconds at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
Time to Maximum Concentration [T(max)] of PBI-200 | 7 days
  Tmax will be determined from the observed plasma concentration data.
Area Under the Concentration-Time Curve (AUC) of PBI-200 from time zero to the time of the last measurable concentration [AUC(0-t)] | 7 days
  AUC, calculated using linear up/ log down trapezoidal method from time zero to time t, where t is the time of the last measurable concentration.
AUC of PBI-200 from time zero to infinity [AUC(0-inf)] | 7 days
  AUC from time zero to infinity, AUC(0-inf) = AUC(0-t) + Ct/ kel, where kel is the terminal rate constant and Ct is the last measurable concentration.

SECONDARY OUTCOMES:
Time of the maximum observed drug concentration [T(max)] | 7 days
  Time of the maximum observed drug concentration
Terminal elimination half-life [T(1/2)] | 7 days
  Apparent terminal elimination half-life, calculated as ln(2)/ kel.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Pyramid Biosciences
Locations (1):
- Bio-Kinetic Clinical Applications, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No